CLINICAL TRIAL: NCT03129256
Title: An Exploratory Study of Low-dose Apatinib Combined With S-1 in Patients With Advanced Non-small Cell Lung Cancer
Brief Title: An Exploration of Apatinib Combined With S-1 in Patients With Advanced Non-small Cell Lung Cancer
Acronym: EASE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Changzhou Cancer Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCH001
Record Dates: First submitted 2017-04-17; First posted 2017-04-26 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Non-small Cell Lung Cancer
Keywords: non-small cell lung cancer; Apatinib; S1
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Apatinib & S-1 (Experimental): Apatinib Mesylate tablet combined with S-1 Capsules Apatinib Mesylate tablet 250mg once daily combined with S-1(Tegafur,Gimeracil and Oteracil Potassium Capsules) 40mg~60mg twice daily by mouth, d1-14, repeated every 3 weeks.
  Interventions: Drug: Apatinib Mesylate tablet combined with S-1 capsules

INTERVENTIONS:
Drug: Apatinib Mesylate tablet combined with S-1 capsules — Oral use with low-dose Apatinib combined with S-1 until disease progression
  Other Names: Ai Tan combined with S-1; Apatinib combined with S-1

SUMMARY:
This study is to explore the potential efficacy and safety of low-dose Apatinib combined with S-1 in patients with advanced lung cancer. Patients with advanced NSCLC will be treated with oral apatinib and S-1 after treatment failure of standard regimen.

DETAILED DESCRIPTION:
Apatinib is a tyrosine kinase inhibitor which selectively inhibits the vascular endothelial growth factor receptor-2 (VEGFR-2). The anti-angiogenesis effect of apatinib has been proved in preclinical tests. Phase II study has showed an improvement of progression free survival in pretreated patients. S-1, an oral fluoropyrimidine has considerable effectiveness with mild side effect in patients failed to standard treatments. The purpose of this study is to evaluate the potential efficacy and safety of low-dose Apatinib combined with S-1 in heavily pretreated patients with advanced lung cancer. And to explore the biomarkers of antiangiogenesis therapy and the possible mechanisms of treatment resistance on the basis of next generation sequencing.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed Non-small cell lung cancer
* Patients with extracranial measurable lesions
* Patients with NSCLC failed for standard treatments
* Eastern Cooperative Oncology Group performance status score: 0~2 and life expectancy of more than 3 months
* Major organs functioning properly
* Compliance is good and agreed to cooperate with the survival of follow-up
* Informed consent

Exclusion Criteria:

* Contraindications for investigational agents
* Patients with clinical symptoms of brain metastases or meningeal metastasis
* Tumor invade big vessels or close to big vessels
* Uncontrolled hypertension
* Abnormal coagulation (INR>1.5 or Prothrombin Time>ULN+4, or Activated Partial Thromboplastin Time>1.5 ULN), bleeding tendency or receiving coagulation therapy
* Hemoptysis, more than 2.5ml daily
* Thrombosis in 12 months, including pulmonary thrombosis, stoke, or deep venous thrombosis.
* Myocardial ischemia or infarction more than stage II, cardiac insufficiency.
* Received big surgery, had bone fracture or ulcer in 4 weeks.
* Urine protein≥++, or urine protein in 24 hours≥1.0g

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival(PFS) | 2 years
  PFS is defined as the length of time from random assignment to disease progression or to death resulting from any cause other than the progress.

SECONDARY OUTCOMES:
Overall Survival(OS) | 2 years
  Overall Survival is defined as the length of time from random assignment to death or to last contact.
Objective response rate(ORR) | 2 years
  Objective response rate is defined as the percentage of subjects having achieved confirmed Complete Response + Partial Response according to Response Evaluation Criteria in Solid Tumors 1.1（RECIST1.1）
Disease Control Rate(DCR) | 2 years
  Disease Control Rate is defined as the percentage of subjects having achieved confirmed Complete Response + Partial Response + Stable Disease according to radiological assessments.
Adverse Events(AEs) | 2 years
  AEs are evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events v4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Tong Zhou, Dr., Principal Investigator — Changzhou Cancer Hospital of Soochow University
Locations (1):
- Changzhou Cancer Hospital of Soochow University, Changzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No